CLINICAL TRIAL: NCT07235956
Title: A Study on the Prediction of the Success Rate of Weaning From Invasive Mechanical Ventilation in Patients by the Ratio of Diaphragmatic Mobility Between the Mid-clavicular Line and the Mid-axillary Line
Brief Title: The Ratio of Diaphragmatic Movement Between the Midaxillary Line and the Midclavicular Line Predicts the Success Rate of Weaning From Mechanical Ventilation
Status: Not yet recruiting | Type: Observational
Sponsor: Zheng Qingjiang (Other)
Responsible Party: Sponsor-Investigator, Zheng Qingjiang, Attending, Zhangzhou Municipal Hospital
Organization: Zhangzhou Municipal Hospital (Other)
Other Study IDs: 2025LWB429
Record Dates: First submitted 2025-09-23; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Mechanical Ventilation
Keywords: Diaphragmatic mobility; Invasive mechanical ventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group with successful extubation of invasive mechanical ventilation
  Interventions: Diagnostic Test: Observe the ratio of diaphragmatic excursion between the midaxillary line and the midclavicular line in the successful group of invasive mechanical ventilation weaning.

INTERVENTIONS:
Diagnostic Test: Observe the ratio of diaphragmatic excursion between the midaxillary line and the midclavicular line in the successful group of invasive mechanical ventilation weaning. — Observe the ratio of diaphragmatic excursion between the midaxillary line and the midclavicular line in the successful group of invasive mechanical ventilation weaning.

SUMMARY:
This study will provide individualized objective indicators for patients undergoing invasive mechanical ventilation. It will set specific assessment parameters for weaning and extubation for different patients, increase the success rate of weaning, avoid the damage and medical risks of re-intubation, and shorten the hospital stay. The main observation targets of this study are: whether weaning is successful; the secondary targets are: specific numerical values of diaphragmatic mobility along the midclavicular line and midaxillary line, oxygenation index, and whether re-intubation occurs within 48 hours. This study is an observational study. The expected study duration is 18 months, and there is no risk of study interruption.

DETAILED DESCRIPTION:
Research Background: Invasive mechanical ventilation is a commonly used rescue measure for critically ill patients. After treatment and improvement, due to factors such as disease damage and the patient's physical condition, one-third of the patients will become dependent on ventilators, resulting in failed weaning. The diaphragm, as the most crucial respiratory muscle, undertakes 60-79% of the ventilation function. However, a combination of factors such as invasive mechanical ventilation, analgesic and sedative drugs, muscle relaxants, disease damage, delayed rehabilitation, and insufficient nutrient supply can lead to rapid diaphragm atrophy in patients. Therefore, an objective and accurate assessment of diaphragm function is crucial for predicting the wear-off success rate of patients with invasive mechanical ventilation. It is of great significance. At present, the research on diaphragmatic ultrasound mainly focuses on diaphragmatic mobility, diaphragmatic thickening rate, and peak diaphragmatic contraction. However, there are differences in the basal diaphragmatic thickness and mobility among each patient. Moreover, the physiological contraction amplitudes of the diaphragm are different, such as smaller ventral amplitude and larger dorsal amplitude. Our research measured the diaphragmatic mobility along the midaxillary line and the midclavicular line, and calculated the ratio of the two. Taking the successful weaning of patients as the main criterion, they were divided into the successful weaning group and the failed weaning group. The odds ratios of the two groups were compared for statistical analysis to determine whether there were statistical differences. The purpose was to provide individualized objective parameters for the weaning and extubation of patients with invasive mechanical ventilation.

Research Objective: This study aims to provide individualized objective indicators for patients on invasive mechanical ventilation, assess parameters for weaning and extubation for different patients, increase the success rate of weaning, avoid the injury and medical risks of re-intubation within 48 hours, and shorten the hospital stay. The primary observation objective of this study is whether weaning is successful or not. The secondary objectives are the specific values of diaphragmatic mobility at the midclavicular and midaxillary lines, oxygenation index, and whether re-intubation occurs within 48 hours. This study is an observational study, with an expected research period of 18 months, and there is no risk of study interruption.

This study is an observational cohort study. Patients who received invasive mechanical ventilation in the intensive care unit of our hospital from October 1, 2025 to December 31, 2026 were collected. The diaphragmatic excursion at the midclavicular line and the midaxillary line of each patient was measured using ultrasound, and the ratio of the diaphragmatic excursion of the two was calculated. The main content was to monitor the diaphragmatic excursion at the midclavicular line and the midaxillary line, and calculate the ratio; the monitoring time points were the first day, the third day, the seventh day (if applicable), the 14th day (if applicable), and before weaning and extubation, while observing the patients' serum albumin, serum prealbumin, hemoglobin, oxygenation index, etc. for treatment. The research content only focuses on human samples and medical treatment data, not on research interventions on the human body.

Research Design: This study is a retrospective observational case-control study. Based on: By reviewing previous literature and using the formula for calculating sample size in medicine: n = Z² × σ²/d² (where, Z is the confidence interval, n is the sample size, d is the sampling error range, σ is the standard deviation, typically taken as 0.5), the sample size was calculated to be 120 cases. According to whether the weaning was successful or not, the cases were divided into the successful group and the failed group; the parameters such as the ratio of diaphragm movement, PA, aPA, oxygenation index at the above time points were collected between the two groups for statistical analysis; the data were analyzed using SPSS 25.0 version (IBM Company, Armonk, New York, USA). The Shapiro-Wilk test was used to evaluate the normality of continuous variables. Variables with normal distribution were presented in the form of mean ± standard deviation and compared using the Student t-test. Variables with non-normal distribution were presented in the form of median (interquartile range) and compared using the Mann-Whitney U test. Categorical variables were presented in the form of frequency (percentage) and compared using the chi-square test or Fisher's exact test. In pairwise comparisons of ultrasound parameters at different time points within each group, repeated measures analysis of variance with Bonferroni correction was used. The receiver operating characteristic (ROC) curve was constructed to evaluate the predictive value of ultrasound parameters for 28-day mortality. The area under the curve (AUC) was calculated, and the optimal cut-off value was determined using the Youden index. A bilateral p-value < 0.05 is considered statistically significant. To address potential confounding factors, a multivariate logistic regression analysis was conducted, and age and the Acute Physiology and Chronic Health Evaluation II score (APACHE II) were adjusted simultaneously.

ELIGIBILITY:
Inclusion Criteria:

Patients who were admitted to the ICU and had invasive mechanical ventilation for more than 72 hours.

Exclusion Criteria:

Patients with irreversible multi-organ failure; Patients with advanced tumors

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is an observational cohort study. Patients who received invasive mechanical ventilation in the intensive care unit of our hospital from October 1, 2025 to December 31, 2026 were collected. The diaphragmatic excursion at the midclavicular line and the midaxillary line of each patient was measured using ultrasound, and the ratio of the diaphragmatic excursion at the two lines was calculated. The main content was to monitor the diaphragmatic excursion at the midclavicular line and the midaxillary line, and calculate the ratio; the monitoring time points were the first day, the third day, the seventh day (if applicable), the 14th day (if applicable), and before weaning and extubation, and at the same time, the patients' serum albumin, serum prealbumin, hemoglobin, oxygenation index, etc. were observed for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of weaning from invasive mechanical ventilation | From enrollment to the outcome of extubation with invasive mechanical ventilation

IPD SHARING:
Plan to Share IPD: No
We have signed a personal informed consent form with the patient, and the patient's private information is protected from disclosure.